CLINICAL TRIAL: NCT05643638
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Phase II Study to Investigate the Efficacy and Safety of CYP-001 in Combination With Corticosteroids vs Corticosteroids Alone for the Treatment of High-Risk Acute Graft Versus Host Disease
Brief Title: A Study of CYP-001 in Combination With Corticosteroids in Adults With High-risk aGvHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cynata Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYP-GvHD-P2-01
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease, Acute
MeSH Terms: conditions — Graft vs Host Disease | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYP-001 plus corticosteroids (Experimental)
  Interventions: Biological: CYP-001: Cymerus induced pluripotent stem cell (iPSC)-derived mesenchymal stem cells (MSCs); Drug: Corticosteroids
- Placebo plus corticosteroids (Placebo Comparator)
  Interventions: Biological: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Biological: CYP-001: Cymerus induced pluripotent stem cell (iPSC)-derived mesenchymal stem cells (MSCs) — Cymerus MSCs are derived from iPSCs using the proprietary Cymerus platform technology.
  Arms: CYP-001 plus corticosteroids
Biological: Placebo — The placebo product is identical to CYP-001, except that it contains no active agent
  Arms: Placebo plus corticosteroids
Drug: Corticosteroids — All enrolled subjects in this trial must receive corticosteroids at a minimum dose of oral prednisone 2 mg/kg/day (or methylprednisolone 1.6 mg/kg/day IV) as therapy for aGvHD for at least for 72 hours post enrollment.

SUMMARY:
This study is a prospective randomized placebo-controlled phase 2 study to compare CYP-001 plus corticosteroids (CS) to placebo plus CS in allogeneic hematologic stem cell transplant recipients with HR-aGvHD. Severity of GvHD will be assessed at screening and throughout the study using Mount Sinai Acute GvHD International Consortium (MAGIC) guidelines. Eligible subjects will be randomized to receive either CYP-001 IV infusion on Days 0 and 4 or placebo on the same days. All subjects will receive ongoing CS therapy as appropriate per institutional guidelines. Subjects will have study visits up to Day 100 during the Primary Evaluation Period. During the Follow-Up Period, subjects will have study visits up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Undergone allogeneic hematopoietic stem cell transplant (HSCT)
* Clinically diagnosed with acute GvHD requiring systemic therapy with corticosteroids.
* HR-aGvHD must meet one of the following clinical features within 72 hours prior to randomization: (a) high-risk as per Refined Minnesota Criteria; OR (b) One of the following: (i) isolated stage 2 involvement of the lower GI tract; (ii) Stage 1 lower GI tract disease with skin involvement
* Evidence of myeloid engraftment post allogeneic HSCT
* Life expectancy of at least one month

Exclusion Criteria:

* Received any systemic treatment for aGvHD other than corticosteroids +/- calcineurin inhibitors
* Chronic GvHD or overlap syndrome with both acute and chronic features of GvHD
* Relapsed primary malignancy since
* received more than one allogeneic HSCT
* Clinically significant respiratory, renal or cardiac disease
* Cholestatic disorders or sinusoidal obstructive syndrome/veno-occlusive disease of the liver
* Any active uncontrolled infection requiring treatment and likely to impact on the ability of the subject to participate in the trial.
* Known infection with CMV, EBV, HHV-6, HBV, HCV, HIV or Tuberculosis. If the treatment for CMV, EBV, HHV-6, HBV, HCV has commenced the subject is eligible.
* Known sensitivity to dimethylsulfoxide (DMSO) or any other component of CYP-001.
* Received any investigational treatment agent within 30 days or within 5 half-lives of Screening, whichever is greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 28 days
  ORR is defined as the proportion of subjects demonstrating a complete response (CR) or partial response (PR) without requirement for additional systemic therapies for an earlier progression, a mixed response or a nonresponse.

SECONDARY OUTCOMES:
Durable Overall response rate (ORR) | 100 days
  Durable ORR is defined as the proportion of subjects demonstrating OR at Day 28 and maintaining OR at Day 60 and Day 100
Overall response rate (ORR) | 100 days
  ORR is defined as the proportion of subjects demonstrating a CR or PR without requirement for additional systemic therapies for an earlier progression, a mixed response or a nonresponse.
Complete response rate (CRR) | 100 days
  ORR is defined as the proportion of subjects demonstrating a CR without requirement for additional systemic therapies for an earlier progression, a mixed response or a nonresponse.
Overall survival | 2 years
  The Kaplan Meier curve will be used to estimate the distribution of overall survival and the probability of surviving to relevant timepoints.
Event-free survival | 2 years
  Event-Free survival is defined as the time from the date of randomization to the date of hematologic disease relapse/progression, graft failure, or death due to any cause.
Time to non-relapse mortality | 2 years
  Time to non-relapse mortality is defined as the time from the date of randomization to the date of death not preceded by hematologic disease relapse/progression.
Failure-free survival | 2 years
  Failure-free survival is defined as the time from the date of randomization to date of hematologic disease relapse/progression, non-relapse mortality, or addition of new systemic aGvHD treatment
Time to malignancy relapse/progression | 2 years
  Time to malignancy relapse/progression is defined as the time from the date of randomization to the date to hematologic malignancy relapse/progression.
Incidence of chronic GvHD | 2 years
  Chronic GvHD is defined as the diagnosis of mild, moderate, or severe chronic GvHD.
Weekly cumulative steroid dose | 100 days
  The total corticosteroid dose administered each week
Patient reported outcomes: Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT) instrument | 2 years
  The FACT-BMT form was designed to measure the quality of life in patients undergoing bone marrow transplantation.
Patient reported outcomes: EuroQol 5-Dimension (EQ-5D) health-related quality of life instrument | 2 years
  EQ-5D is a standardized measure of health-related quality of life
Incidence, severity, duration of treatment-emergent adverse events | 2 years
  Assessment of safety

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Airey, MD, Study Director — Cynata Therapeutics Limited
Locations (39):
- United States (13):
  - Banner MD Anderson, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Memorial healthcare System, Pembroke Pines, Florida
  - BMT Group of Georgia, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - University Of Nebrasaka Medical Center, Omaha, Nebraska
  - Weill Cornell Medicine - New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
- France (3):
  - Hospital Claude Huriez, Lille
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
- Italy (6):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale dell'Angelo di Mestre, Venezia
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Spain (6):
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitato De La Princesa, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clínica Universidad de Navarra, Pamplona
- Turkey (Türkiye) (7):
  - Anadolu Medical Center, Eskişehir
  - Gayrettepe Florence Nightingale Hastanesi, Istanbul
  - Koc University, Istanbul
  - Memorial Bahcelievler Hospital, Istanbul
  - Izmir Medicalpark Hospital, Izmir
  - İnonu University, Malatya
  - Dr Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Yenimahalle

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will consider requests to share IPD from this study for further research of a non-commercial nature. Requests should be submitted to clinical@cynata.com. Sharing of IPD will be subjects to the execution of an IPD sharing agreement, and applicable laws, regulations and guidance in force at that time.
Time Frame: IPD sharing requests will be considered from 12 months after publication of results of this study.
Access Criteria: Requests for sharing of IPD for non-commercial research purposes will be considered in good faith by the Sponsor. Requests must be accompanied by a detailed research plan, with a justification for the proposed research.